CLINICAL TRIAL: NCT01217645
Title: A Phase I, Open-label, Single-Centre Study to Assess the Distribution, Metabolism and Excretion of [14C]AZD6765 After a Single-Dose Intravenous Administration to Healthy Male Subjects
Brief Title: Study to Assess the Distribution, Metabolism and Excretion of [14C]AZD6765 After a Single-Dose Intravenous Administration
Acronym: AZD6765
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D6702C00030
Record Dates: First submitted 2010-07-29; First posted 2010-10-08 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Major Depressive Disorder
Keywords: Major depression disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — AZD6765

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 150 mg [14C] AZD6765 (Experimental)
  Interventions: Radiation: 150 mg [14C] AZD6765

INTERVENTIONS:
Radiation: 150 mg [14C] AZD6765

SUMMARY:
This is a study to assess the distribution, metabolism and excretion of [14C]AZD6765 after a single-dose intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a normal creatinine clearance of ≥60 mL/min
* Subjects who self-identify their race as Asian

Exclusion Criteria:

* History of any clinically significant medical, neurologic or psychiatric disease as judged by the investigator
* History of symptomatic orthostatic hypotension (ie, postural syncope)
* Subjects who have received any radiolabelled study drug within 12 months of the Screening Visit.
* Subjects who are monitored for radioactivity as part of their occupation
* Subjects who have been exposed to radiation levels above background, (eg, throughX-Ray examinations) of >5mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1mSv per year of life.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The change in distribution, metabolism, and elimination of AZD6765 and total radioactivity after single-dose (150 mg) intravenous administration of [14C]-labelled AZD6765 | Blood samples will be taken from predose until upto 240 hrs from start of infusion to assess radioactivity
The change in excretion of 14C (mass balance) in urine and faeces after a single intravenous dose of 150 mg [14C] AZD6765 | Urine and feacal samples will be taken from predose until up to 240 hrs from start of infusion to assess radioactivity

SECONDARY OUTCOMES:
To identify and profile the metabolites in selected samples of urine, faeces and plasma following a single intravenous dose of 150 mg [14C] AZD6765 | A Range from predose until up to 240 hrs from start of infusion.
Safety and tolerability after a single IV administration of [14C] AZD6765 by assessing a panel of measures: adverse events, blood pressure and pulse, blood samples, urinalysis, hematology, clinical chem, physical exam, ECG and symptoms of suicidality. | A Range from predose until up to 240 hrs from start of infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: D6702C00030 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=574&filename=D6702C00030_Clinical_Study_Report_Synopsis.pdf